CLINICAL TRIAL: NCT03833518
Title: Cortical Biomarkers of Hand Function and Recovery After Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We only enrolled one participant, and this participant was withdrawn prior to collecting any useful data. Then, COVID. Now, Dr. Collinger's faculty tenure with the VA ended.
Sponsor: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jennifer Collinger, Research Biomedical Engineer, VA Pittsburgh Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00002855
Record Dates: First submitted 2019-02-04; First posted 2019-02-07 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Stroke; Spinal Cord Injuries
Keywords: hand; rehabilitation; motor cortex
MeSH Terms: conditions — Stroke; Spinal Cord Injuries | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This is a pilot study to collect data to support a VA grant submission to study fMRI and neurophysiological predictors of hand function and recovery during a robotic intervention in people with hand impairments due to stroke or spinal cord injury.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hand impairment due to stroke or spinal cord injury (Experimental): Individuals who have experienced a sub-cortical stroke or a cervical spinal cord injury resulting in loss of hand function.
  Interventions: Other: Rehabilitation using motorized glove for stroke and spinal cord injury; Other: Functional MRI for stroke and spinal cord injury; Other: Transcranial magnetic stimulation (TMS) for stroke and spinal cord injury

INTERVENTIONS:
Other: Rehabilitation using motorized glove for stroke and spinal cord injury — Individuals with hand impairment due to stroke or spinal cord injury will wear a motorized glove (Gloreha Sinfonia), or exoskeleton, as part of a rehabilitation protocol to improve dexterity. For each exercise, participants will attempt to do the action, receiving assistance as necessary via powered motors that can move each finger through its passive range of motion based on the current and target position.
  Other Names: Exoskeleton therapy
Other: Functional MRI for stroke and spinal cord injury — All participants will undergo 3 functional MRI's (fMRI's), two at the beginning of the experiment to document brain activity related to movement intention and ability to sense movement. A third MRI will be performed after the rehabilitation is completed to document the change in brain activity related to movement intention and ability to sense movement.
  Other Names: fMRI
Other: Transcranial magnetic stimulation (TMS) for stroke and spinal cord injury — Stimulation of the nervous system may be performed using a magnetic stimulator. TMS of the central nervous system is optional. Whether or not a participant undergoes TMS will depend upon their consent, their eligibility for TMS (i.e. no seizure history), and their neurological response to TMS.
  Other Names: TMS

SUMMARY:
This is a pilot study to collect data to support a VA grant submission to study fMRI and neurophysiological predictors of hand function and recovery during a robotic intervention in people with hand impairments due to stroke or spinal cord injury.

DETAILED DESCRIPTION:
The loss of arm and hand function after cervical spinal cord injury (SCI) limits independence and increases the cost of care. As a result, Veterans with tetraplegia prioritize restoration of hand and arm function over all other rehabilitation goals. Similar to SCI, stroke of supraspinal areas involved in motor control results in acute movement deficits in more than 85% of survivors. Despite advances in treatment and rehabilitation, 50% of stroke survivors have persistent hand impairment. The loss of hand function and dexterity limits the ability to perform many activities of daily living, and thus limits independence. Since motor deficits are often permanent after SCI and stroke, new strategies are needed to restore dexterous hand function.

Advances in functional imaging have enabled the measurement of finger-related activation patterns in somatosensory cortex, but little is known about how these representational patterns are impacted when hand function is lost. Prior studies of gross movements have reported reorganization of cortical activity after injury. The investigators aim to improve dexterous hand function by increasing our understanding of finger-related cortical reorganization after lesions to the spinal or supraspinal structures. This understanding could allow discrimination between adaptive and maladaptive patterns underlying hand function and guide restorative therapies. Additionally, imaging biomarkers of injury often track with functional recovery.

The aim is to improve dexterous hand function by increasing our understanding of finger-related cortical reorganization after lesions to the spinal or supraspinal structures. This understanding could allow discrimination between adaptive and maladaptive patterns underlying hand function and guide restorative therapies. Additionally, imaging biomarkers of injury often track with functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* Normal or corrected to normal vision
* Hand impairment due to spinal cord injury or stroke
* Weakness of fingers
* One year after stroke or spinal cord injury
* Some proprioception (can feel when finger is moved, without seeing)
* Minimal spasticity

Exclusion Criteria:

* Implanted metal with is unsafe for MRI
* Pregnant or expecting to become pregnant
* History of hand surgery which is under evaluation
* Cognitive or language issues that would interfere with following directions
* Other neurological disorder that would affect movement
* History of seizure or epilepsy
* Body weight > 300 pounds

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Number of participants that show significant finger-specific activation prior to the intervention | Baseline, prior to intervention, week 1
  The investigators will use functional magnetic resonance imaging (fMRI) to measure cortical activity relating to finger-specific brain activation before the rehabilitation intervention.

SECONDARY OUTCOMES:
Change from baseline finger strength after rehabilitation intervention | After intervention, 12 weeks
  The investigators will assess finger strength of participants both before and after the rehabilitation intervention. The change in in finger strength will serve as a secondary outcome measure.
Change from baseline in finger dexterity after rehabilitation intervention | After intervention, 12 weeks
  The investigators will assess each participant's ability to isolate movement of individual fingers both before and after the rehabilitation intervention. The change in this measure of dexterity will serve as a secondary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Collinger, PhD, Principal Investigator — US Department of Veterans Affairs
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Research information will not be shared with anyone outside of the research team.

REFERENCES:
- [Background] Rathore SS, Hinn AR, Cooper LS, Tyroler HA, Rosamond WD. Characterization of incident stroke signs and symptoms: findings from the atherosclerosis risk in communities study. Stroke. 2002 Nov;33(11):2718-21. doi: 10.1161/01.str.0000035286.87503.31. PMID 12411667
- [Background] Peckham PH, Keith MW, Kilgore KL, Grill JH, Wuolle KS, Thrope GB, Gorman P, Hobby J, Mulcahey MJ, Carroll S, Hentz VR, Wiegner A; Implantable Neuroprosthesis Research Group. Efficacy of an implanted neuroprosthesis for restoring hand grasp in tetraplegia: a multicenter study. Arch Phys Med Rehabil. 2001 Oct;82(10):1380-8. doi: 10.1053/apmr.2001.25910. PMID 11588741
- [Background] Anderson KD. Targeting recovery: priorities of the spinal cord-injured population. J Neurotrauma. 2004 Oct;21(10):1371-83. doi: 10.1089/neu.2004.21.1371. PMID 15672628
- [Background] Doll U, Maurer-Burkhard B, Spahn B, Fromm B. Functional hand development in tetraplegia. Spinal Cord. 1998 Dec;36(12):818-21. doi: 10.1038/sj.sc.3100706. PMID 9881729
- [Background] Fawcett JW. Recovery from spinal cord injury: regeneration, plasticity and rehabilitation. Brain. 2009 Jun;132(Pt 6):1417-8. doi: 10.1093/brain/awp121. Epub 2009 May 8. No abstract available. PMID 19429905
- [Background] Nowak DA. The impact of stroke on the performance of grasping: usefulness of kinetic and kinematic motion analysis. Neurosci Biobehav Rev. 2008 Oct;32(8):1439-50. doi: 10.1016/j.neubiorev.2008.05.021. Epub 2008 May 23. PMID 18582943
- [Background] Raghavan P, Petra E, Krakauer JW, Gordon AM. Patterns of impairment in digit independence after subcortical stroke. J Neurophysiol. 2006 Jan;95(1):369-78. doi: 10.1152/jn.00873.2005. Epub 2005 Oct 5. PMID 16207778
- [Background] Lang CE, Schieber MH. Differential impairment of individuated finger movements in humans after damage to the motor cortex or the corticospinal tract. J Neurophysiol. 2003 Aug;90(2):1160-70. doi: 10.1152/jn.00130.2003. Epub 2003 Mar 26. PMID 12660350
- [Background] Lang CE, Schieber MH. Reduced muscle selectivity during individuated finger movements in humans after damage to the motor cortex or corticospinal tract. J Neurophysiol. 2004 Apr;91(4):1722-33. doi: 10.1152/jn.00805.2003. Epub 2003 Dec 10. PMID 14668295
- [Background] Wenzelburger R, Kopper F, Frenzel A, Stolze H, Klebe S, Brossmann A, Kuhtz-Buschbeck J, Golge M, Illert M, Deuschl G. Hand coordination following capsular stroke. Brain. 2005 Jan;128(Pt 1):64-74. doi: 10.1093/brain/awh317. Epub 2004 Oct 7. PMID 15471902